CLINICAL TRIAL: NCT03261518
Title: Investigation of Relationship Between Contrast Nephropathy and Caval Index Measurement in Patients With Suspected Ileus in Emergency Department
Brief Title: Investigation of Relationship Between Contrast Nephropathy and Caval Index Measurement in Patients With Ileus in ED
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Yusuf Uyanik, EMERGENCY MEDICINE RESIDENT, Derince Training and Research Hospital
Other Study IDs: KÜ GOKAEK 2017/1.13
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Ileus; Mechanical; Contrast-induced Nephropathy
Keywords: ileus; Contrast-induced Nephropathy; vena cava inferior
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: inferior vena cava ultrasound — Place the patient in the supine position. The degree of elevation of the head of the bed has not been shown to make a significant difference in measurements. The diameter of the IVC for calculation of the caval index should be measured 2 cm from where it enters the right atrium .An alternative way to visualize respiratory variation is to use M-mode, with the beam overlying the IVC 2 cm from the right atrium.The inspiratory and expiratory diameter can then be measured on the M-mode image, at the smallest and largest locations, respectively.

SUMMARY:
In this study, the investigators aimed to evaluate the incidence of vena cava inferior diamater on ultrasound guidance of intravascular volume before diagnosis of contrast

- enhanced CT for diagnostic purposes in ileus patients and to investigate the incidence and risk of developing contrast nephropathy due to contrast - enhanced CT.

DETAILED DESCRIPTION:
Our work will be carried out in Kocaeli Derince Education and Research Hospital Emergency Service. Patients who are scheduled to receive abdominal contrast computed tomography (CT) scans in the emergency room, who are over 18 years of age, who are referred to Kocaeli Derince Education and Research Hospital Emergency Department for the study, will be calculated and recorded. The Mehran risk scores will be calculated and recorded in our clinic. 3 ml / kg IV physiological saline (SF) is applied first and then 1 ml / kg / hr IV SF is applied for at least 6 hours after shots. In addition, patients with contrasted abdominal CT underwent emergency surveillance ultrasound imaging (including the measurement of the vena cava diameter for evaluation of the patient's volume status). Patients who were admitted to our general surgery and not followed up for at least 48 hours, patients with contrast allergies, patients with renal replacement therapy, pregnancies, patients with contrast-enhanced CT scans within the last 10 days, and patients not informed will not be taken to the study. All Emergency Physicians will be informed about the study. Less than 100 mL of hypoosmolar, non-ionic contrast material will be used for all CT shots. Patients will be evaluated for the development of contrast nephropathy according to biochemical assays 48-72 hours after CT acquisition. Physicians evaluating patients in the emergency and general surgery services will be required to record blood tests that they consider necessary for diagnostic and therapeutic purposes, and no extra blood will be collected for use in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent contrast abdominal CT and were admitted to our general surgery department for at least 48 hours
* Written informed patients
* Patients older than 18 years

Exclusion Criteria:

* With contrast agent allergy
* Story of renal replacement therapy
* Contrast agent exposure within the last 10 days
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-08-24 (Estimated); Primary Completion 2017-12-15 (Estimated); Study Completion 2017-12-15 (Estimated)

PRIMARY OUTCOMES:
Estimate contrast nephropathy in patients with low volume status by calculating Vena cava index | 48 hours
  Estimate contrast nephropathy in patients with low volume status by calculating Vena cava index In this study, we aimed to evaluate the incidence of vena cava inferior vena cava on ultrasound guidance of intravascular volume before diagnosis of contrast-enhanced CT and to investigate the incidence and development of contrast nephropathy due to contrast-enhanced CT.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Habeb M, Agac MT, Aliyev F, Pehlivanoglu S, Ongen Z. [Contrast media-induced nephropathy: clinical burden and current attempts for prevention]. Anadolu Kardiyol Derg. 2005 Jun;5(2):124-9. Turkish. PMID 15939688
- [Background] McCullough PA, Choi JP, Feghali GA, Schussler JM, Stoler RM, Vallabahn RC, Mehta A. Contrast-Induced Acute Kidney Injury. J Am Coll Cardiol. 2016 Sep 27;68(13):1465-1473. doi: 10.1016/j.jacc.2016.05.099. PMID 27659469
- [Background] Sanaei-Ardekani M, Movahed MR, Movafagh S, Ghahramani N. Contrast-induced nephropathy: a review. Cardiovasc Revasc Med. 2005 Apr-Jun;6(2):82-8. doi: 10.1016/j.carrev.2005.07.004. PMID 16263365
- [Background] Kelly AM, Dwamena B, Cronin P, Bernstein SJ, Carlos RC. Meta-analysis: effectiveness of drugs for preventing contrast-induced nephropathy. Ann Intern Med. 2008 Feb 19;148(4):284-94. doi: 10.7326/0003-4819-148-4-200802190-00007. PMID 18283206